CLINICAL TRIAL: NCT07400510
Title: Improving Lower Extremity DVT Outcomes in the Outpatient Setting: An Evaluation of 3-Point of Care Ultrasound for Timely Diagnosis and Treatment
Brief Title: DVT Evaluation Using POCUS for Diagnosis and Treatment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Stephanie A. Carey, MD, Assistant Professor of Family & Community Medicine, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00027831
Record Dates: First submitted 2026-01-28; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Deep Venous Thromboses
Keywords: POCUS; DVT; Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- POCUS positive, High risk, STAT DVT (Experimental): Patient who is high risk for DVT had a positive POCUS study in office was referred for STAT DVT study.
  Interventions: Diagnostic Test: STAT Venous Duplex
- POCUS positive, Low risk, STAT DVT (Experimental): Patient who is low risk for DVT had a positive POCUS study in office was referred for STAT DVT study.
  Interventions: Diagnostic Test: STAT Venous Duplex
- POCUS negative, High risk, STAT DVT (Experimental): Patient who is high risk for DVT had a negative POCUS study in office was referred for STAT DVT study.
  Interventions: Diagnostic Test: STAT Venous Duplex
- POCUS negative, Low risk, Routine DVT (Experimental): Patient who is low risk for DVT had a negative POCUS study in office was referred for routine DVT study.
  Interventions: Diagnostic Test: Routine Venous Duplex

INTERVENTIONS:
Diagnostic Test: STAT Venous Duplex — STAT Venous Duplex
  Arms: POCUS negative, High risk, STAT DVT; POCUS positive, High risk, STAT DVT; POCUS positive, Low risk, STAT DVT
Diagnostic Test: Routine Venous Duplex — Routine Venous Duplex
  Arms: POCUS negative, Low risk, Routine DVT

SUMMARY:
This study will include approximately 50 patients who will be enrolled if there is suspicion of lower extremity deep vein thrombosis (DVT). Each patient will receive a point-of-care ultrasound performed by physicians in an outpatient clinic. All patients will receive a subsequent confirmatory gold standard venous duplex ultrasonography. The investigators will compare time to diagnosis and treatment initiation and evaluate short-term clinical outcomes, including pulmonary embolism, hospitalization, ICU care, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Penn State health patient
* 18 years and older
* English speaking
* Presentation at clinical office with symptoms of a DVT

Exclusion Criteria:

* Pregnancy
* Less than 18 years old
* Non-English speaking
* Chronic Deep Vein Thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects Who Have Identical POCUS Result to Venous Duplex Result | 1 week
  Number of subjects whose ultrasound results using POCUS and subsequent confirmatory gold standard venous duplex ultrasound are identical, whether positive or negative for DVT.

SECONDARY OUTCOMES:
Rate of Pulmonary Embolism | 3 months
  Rate of morbidity will be monitored for 3 months following the diagnosis of DVT by confirmatory venous duplex. Rate of morbidity will be identified through emergency room visits related to the DVT and hospitalizations related to the DVT.
Rate of Stroke | 3 months
  Rate of morbidity will be monitored for 3 months following the diagnosis of DVT by confirmatory venous duplex. Rate of morbidity will be identified through emergency room visits related to the DVT and hospitalizations related to the DVT.
Rate of Myocardial Infarction | 3 months
  Rate of morbidity will be monitored for 3 months following the diagnosis of DVT by confirmatory venous duplex. Rate of morbidity will be identified through emergency room visits related to the DVT and hospitalizations related to the DVT.
Number of Subjects who Died | 3 months
  Number of subjects who died will be monitored for 3 months following the diagnosis of DVT by confirmatory venous duplex.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Health, Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided